CLINICAL TRIAL: NCT05236868
Title: An Open-Label, Single-Dose Study to Assess the Absolute Oral Bioavailability and Pharmacokinetics of JNJ-42847922 (Seltorexant) Administered as Oral Tablet and an Intravenous Microdose of 14C-seltorexant in Healthy Participants
Brief Title: A Study of JNJ-42847922 (Seltorexant) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109133; 42847922MDD1019 (Other: Janssen Research & Development, LLC); 2021-004068-92 (EudraCT Number)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Seltorexant (Experimental): Participants will receive a single oral dose of seltorexant. At 2 hours after oral dosing, participants will receive 14C-seltorexant as an intravenous (IV) infusion over 15 minutes.
  Interventions: Drug: Seltorexant

INTERVENTIONS:
Drug: Seltorexant — Seltorexant will be administered orally as a tablet and as an intravenous infusion of 14C-seltorexant.
  Other Names: JNJ-42847922

SUMMARY:
The purpose of this study is to determine the absolute bioavailability of seltorexant in healthy participants following a single oral dose of seltorexant and an intravenous (IV) infusion dose of 14C-seltorexant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history at screening and physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and at admission to the study site on Day 1
* Healthy on the basis of clinical laboratory tests performed at screening and at admission to the study site on Day -1
* All female participants (regardless of childbearing potential), must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1
* A woman must be a) Not of childbearing potential; b) Of childbearing potential and practicing a highly effective method of contraception (failure rate of less than (<) 1 percent (%) per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study intervention and until 3 months after the study treatment administration
* Must sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study site (Day -1) as determined by the investigator. Alanine transaminase (ALT)/aspartate transaminase (AST) concentrations within normal range at screening. One retest for ALT/AST is permitted
* Clinically significant abnormal physical examination, vital signs, or 12-lead (ECG) at screening or at admission to the study site on Day -1 as determined by the investigator
* Participant has a current or recent history of serious suicidal ideation within the past 6 months, corresponding to a positive response on item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) for ideation on the Columbia-Suicide Severity Rating Scale (C SSRS), or a lifetime history of suicidal behavior or suicidal attempt as validated by the C SSRS at screening
* Positive test for human immunodeficiency virus (HIV)-1 and HIV-2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies
* Has any history or current diagnosis of obstructive sleep apnea or parasomnias. Participants with restless leg syndrome/periodic leg movement disorder or insomnia disorder are allowed if not requiring medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Absolute Bioavailability | Up to Day 4
  Absolute bioavailability is calculated as the ratio of dose normalized area under the plasma drug concentration-time curve (AUC) of oral and intravenous (IV) administration.

SECONDARY OUTCOMES:
Area Under the Plasma Analyte Concentration Versus Time Curve of Seltorexant from Time Zero to Infinite time (AUC [0-Infinity]) | Up to Day 4
  AUC (0-infinity) is defined as the area under the plasma analyte concentration versus time curve of seltorexant from time zero to infinite time.
Area Under the Plasma Analyte Concentration Versus Time Curve of Seltorexant from Time Zero to Time of the Last Measurable Concentration (AUC [0-Last]) | Up to Day 4
  AUC (0-Last) is defined as area under the plasma analyte concentration versus time curve from time zero to time of the last measurable (non- below quantifiable limit [BQL]) concentration.
Maximum Observed Plasma Analyte Concentration (Cmax) of Seltorexant | Up to Day 4
  Cmax of Seltorexant will be reported.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Seltorexant | Up to Day 4
  Tmax of Seltorexant will be reported.
Apparent Terminal Elimination Half-life (t1/2) of Seltorexant | Up to Day 4
  Apparent terminal elimination half-life is calculated as 0.693/ lambda(z).
Number of Participants with Adverse Events (AEs) | Screening (up to -21 days) up to Day 7
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency